CLINICAL TRIAL: NCT01152528
Title: VA-SENSE - BACTERIAL VAGINOSIS ONCE A WEEK SCREENING AND TREATMENT TO REDUCE INFECTIVE COMPLICATIONS, ABORTION AND PRETERM DELIVERY IN PREGNANT WOMEN WITH PREVIOUS PRETERM DELIVERY.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Common Sense (Other)
Responsible Party: Hadar Kessary, Common Sense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: F-7-27.3-1
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Vaginal Infections; Bacterial Vaginosis; Late Miscarriage; Preterm Birth; Preterm Premature Rupture of Membranes
Keywords: bacterial vaginosis; screening; abortion; preterm delivery
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Premature Birth; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VA-SENSE — The VA-SENSE contains a strip of pH indicator (color indicator) that is sensitive to the acidity level. A change in the color of the strip due to changes in the acidity level of vaginal secretions absorbed in the panty liner clearly indicates high probability of bacterial or parasitic vaginal infection. Any color change that results from contact with urine will disappear 10 minutes of drying out, and then the color of the indicator strip will fade back to the original color (yellow).

SUMMARY:
The purpose of this study is to determine whether screening of pregnant women with history of previous preterm delivery, once a week, for bacterial vaginosis using VA-SENSE, and treatment of positive women will reduce the risk of spontaneous preterm birth. We will compare between the effectiveness of once a week screening and once during pregnancy screening.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant subjects, aged 18-50 years, pregnancy week 10 or less or 20 or less, with history of previous preterm delivery.
2. Subject is ready to sign an informed consent form.

Exclusion Criteria:

1. Subject with ruptured membranes.
2. Subject with signs and symptoms of bacterial vaginosis or Trichomoniasis infections.
3. Subject with blood in her vaginal secretions.
4. Subject is currently participating in another clinical study.
5. Subject is unable or unwilling to cooperate with study procedures.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth, gestational week at delivery. | 9 months
  Each participant will use at least 8 VA-SENSE (maximum 20 TPLs), once a week for at least 8 weeks (maximum 20 weeks), or will be screened by VS-SENSE once during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Western Galilee, Israel